CLINICAL TRIAL: NCT06576882
Title: 7-day Versus 14-day Vonoprazan-based Triple Therapy for Eradication of H. Pylori in Adolescents: A Randomized Controlled Trial
Brief Title: 7 Days vs. 14 Days of Vonoprazan-based Triple Therapy for H. Pylori Eradication
Acronym: VOTE-HP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sameh A. Lashen, Assistant Professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0306630
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-04

CONDITIONS: Helicobacter Pylori Infection; Gastritis; Vonoprazan; Adolescents
Keywords: Helicobacter pylori; Vonoprazan; Triple therapy; Adolescent; Eradication rate; Children
MeSH Terms: conditions — Gastritis | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Clarithromycin

STUDY DESIGN:
Intervention Model Description: 1:1 assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 14-days Vonoprazan-based triple therapy (Active Comparator): Vonoprazan tablets 20 mg twice daily plus Amoxicillin 50 mg/kg/day capsules or suspension [maximum daily dose 2 g] plus Clarithromycin 20 mg/kg/day tablets or suspension [maximum daily dose 1 g]. The triple combination will be given for 14 days .
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Clarithromycin
- 7-days Vonoprazan-based triple therapy (Experimental): Vonoprazan tablets 20 mg twice daily plus Amoxicillin 50 mg/kg/day capsules or suspension [maximum daily dose 2 g] plus Clarithromycin 20 mg/kg/day tablets or suspension [maximum daily dose 1 g]. The triple combination will be given for 7 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Clarithromycin

INTERVENTIONS:
Drug: Vonoprazan — Participants will receive Vonoprazan 20 mg tablets twice daily before meals.
  Other Names: Vonacidan; Tavoniza; Vondalous; Vonaspire; Vonseca
Drug: Amoxicillin — Participants will receive Amoxicillin 50 mg/kg/day capsules or suspension [maximum daily dose: 2 g].
  Other Names: Emox; Ibiamox; Amoxicid
Drug: Clarithromycin — Participants will receive Clarithromycin 20 mg/kg/day tablets or suspension [maximum daily dose: 1 g].
  Other Names: Klacid; Klarithro; Klarimix; Infectocure

SUMMARY:
The study aims to test the efficacy of 7 days vs. 14 days of Vonoprazan-triple therapy in the eradication of Helicobacter Pylori infection in adolescents and young children.

DETAILED DESCRIPTION:
After being informed about the study details, all eligible participants (or their legal guardians) will give informed written consent to be involved. After a one week screening, eligible participants will be randomized to Vonoprazan plus Amoxicillin plus Clarithromycin triple therapy for either 14 days (group 1), or 7 days (group 2) at a 1:1 ratio. After the end of therapy, H. Pylori eradication will be evaluated after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants in the age group (10-18 years), both genders, referred with dyspeptic complaints such as heartburn, dyspepsia, nausea, and epigastric pain who are positive for H. Pylori infection by a standardized diagnostic test.
2. Pediatric patients with a clinical, laboratory, and endoscopic diagnosis of H.P.-positive gastritis and the other conditions necessary for H.P. eradication, according to the Maastricht V consensus report .

Exclusion Criteria:

1. allergy to any of the drugs used in the study
2. previous attempts to eradicate H.P.
3. receipt of antibiotics, PPIs, bismuth, H2 antagonists or probiotics within 4 weeks of the study.
4. Children with the diagnosis of any condition that might affect the absorption of drugs such as celiac disease or Crohn's disease.
5. hepatic impairment or kidney failure.
6. symptoms suggestive of functional disorders.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 326 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
H. Pylori eradication rate | 4 weeks after completion of treatment
  Number of participants who will achieve a negative H. pylori antigen detection test after the end of therapy.

SECONDARY OUTCOMES:
Adverse events during treatment. | From first dose of treatment until 7 or 14 days of treatment regimen assigned.
  Type and frequency of treatment-related adverse effects in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Sameh A Lashen, MD, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria University., Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Clinico-laboratory data can be shared, but participant-specific identity data cannot be shared to maintain participant confidentiality.